CLINICAL TRIAL: NCT03304470
Title: A Double-Blind, Randomized, Intraindividual, Vehicle-Controlled, Phase 2 Study to Evaluate the Safety and Efficacy of Topically Applied ATx201 in Subjects With Moderate Atopic Dermatitis
Brief Title: A Study to Evaluate the Safety and Efficacy of ATx201 in Subjects With Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNION therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATx201-003
Record Dates: First submitted 2017-09-25; First posted 2017-10-09 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATx201 2% CREAM (Experimental)
  Interventions: Drug: ATx201 2% Cream
- ATx201 Cream Vehicle (Placebo Comparator)
  Interventions: Drug: ATx201 Cream Vehicle

INTERVENTIONS:
Drug: ATx201 2% Cream — Anhydrous Cream
  Arms: ATx201 2% CREAM
Drug: ATx201 Cream Vehicle — Anhydrous Cream
  Arms: ATx201 Cream Vehicle

SUMMARY:
This is a Phase 2, 3-week, single-center, double-blind, randomized, two-arm, vehicle controlled study, with each individual receiving both active and vehicle treatment. Approximately 30 subjects with moderate atopic dermatitis will receive topically applied ATx201 CREAM 2% and matching vehicle once daily for 3 weeks (5 mg/cm2/day), without occlusion. ATx201 and vehicle will be applied on two separate target lesions of moderate atopic dermatitis (lesions of at least 3 × 3 cm, excluding the face, scalp, genitals, hands, and feet, ideally from the same anatomical location).

ELIGIBILITY:
Inclusion Criteria:

* clinically confirmed diagnosis of active atopic dermatitis
* at least a 6-month history of atopic dermatitis and had no significant flares in atopic dermatitis for at least 4 weeks before screening
* ≥2 areas of atopic dermatitis (excluding face, scalp, genitals, hands, and feet) of at least 3 × 3 cm; with a lesional TSS of ≥5 at Day 1 for each treatment area

Exclusion Criteria:

* breastfeeding, pregnant, or is planning to become pregnant during the study.
* clinically infected atopic dermatitis
* Fitzpatrick's Skin Phototype ≥5
* Presence of any tattoos, scratches, open sores, excessive hair, or skin damages in the target lesion areas
* known to have immune deficiency or is immunocompromised.
* history of cancer or lymphoproliferative disease within 5 years prior to Day 1.
* major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study.
* clinically significant medical condition or physical/laboratory/vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.
* known history of chronic infectious disease (e.g., hepatitis B, hepatitis C, or infection with human immunodeficiency virus).
* used hydroxyzine or diphenhydramine within 1 week prior to Day 1.
* used dupilumab within 12 weeks prior to Day 1.
* received any nonbiological investigational product or device within 4 weeks prior to Day 1
* used crisaborole and any other topical PDE-4 inhibitor within 4 weeks prior to Day 1.
* used doxepin within 1 week prior to Day 1.
* used topical products containing urea within 1 week prior to Day 1.
* used nonurea-containing emollient anywhere on the body from 1 day before Day 1.
* used systemic antibiotics or topical antibiotics on the treated areas within 2 weeks prior to Day 1.
* used any topical medicated treatment for atopic dermatitis within 2 weeks prior to Day 1, including, but not limited to, topical corticosteroids, calcineurin inhibitors, tars, bleach, antimicrobials, medical devices, and bleach baths.
* used systemic treatments (other than biologics) that could affect atopic dermatitis less than 4 weeks prior to Day 1 (e.g., retinoids, calcineurin inhibitors, methotrexate, cyclosporine, hydroxycarbamide [hydroxyurea], azathioprine, oral/injectable corticosteroids).
* received any marketed or investigational biological agent within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
* excessive sun exposure, is planning a trip to a sunny climate, has received ultraviolet phototherapy, or has used tanning booths within 4 weeks prior to Day 1, or is not willing to minimize natural and artificial sunlight exposure during the study. Use of sunscreen products (excluding the treatment areas) and protective apparel are recommended when exposure cannot be avoided.
* known or suspected allergy to ATx201 or any component of the investigational product.
* known history of clinically significant drug or alcohol abuse in the last year prior to Day 1.
* history of an allergic reaction or significant sensitivity to lidocaine or other local anesthetics.
* history of hypertrophic scarring or keloid formation in scars or suture sites.
* taking anticoagulant medication, such as heparin, low molecular weight-heparin, warfarin, or antiplatelets (nonsteroidal anti-inflammatory drugs and aspirin ≤81 mg will not be considered antiplatelets) within 2 weeks prior to Day 1, or has a contraindication to skin biopsies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Incidence of local and systemic treatment-emergent adverse events | 34 days
  # of TEAEs

SECONDARY OUTCOMES:
Change from baseline in lesional Total Sign Score at Days 8, 15, and 22. | 22 Days
Change from baseline in lesional Treatment Areas Assessment at Days 8, 15, and 22 | 22 Days
Change from baseline in skin barrier and biomarker levels at Day 22 | Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Prokocimer, Study Director — Sponsor CMO
Locations (1):
- Innovaderm Research Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No